CLINICAL TRIAL: NCT05817630
Title: Impact of Duration of Silicone Oil Tamponade on Foveal and Parafoveal Thickness in Rhegmatogenous Retinal Detachment: A Retrospective Cohort Study
Brief Title: Duration of Silicone Oil Tamponade on Foveal and Parafoveal Thickness in Rhegmatogenous Retinal Detachment
Acronym: siliconeoil
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, Associate Professor of Ophthalmology Cairo university, Dar El Oyoun Hospital
Other Study IDs: N-19-2023
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group A: 3 months SO Tamponade
  Interventions: Other: Silicone oil Tamponade for Retinal Detachment
- Group B: Group B: 6 months SO Tamponade
  Interventions: Other: Silicone oil Tamponade for Retinal Detachment

INTERVENTIONS:
Other: Silicone oil Tamponade for Retinal Detachment — eyes with Rhegmatogenous Retinal Detachment (RRD, for whom pars plana vitrectomy and silicone oil had been performed

SUMMARY:
Our study observes and analyses the influence of the duration of tamponade with silicone oil on the foveal and parafoveal thickness.

DETAILED DESCRIPTION:
Retrospective Cohort study Retrospective review of records of eyes with Rhegmatogenous Retinal Detachment (RRD, for whom pars plana vitrectomy and silicone oil had been performed, in the period between January 2019 and December 2021.

After checking inclusion and exclusion criteria; we will enroll all the cases.

We shall observe the duration of silicone oil tamponade, and then divide the cases; accordingly; into 2 groups (Cohort).

* Group A: 3 months SO Tamponade
* Group B: 6 months SO Tamponade

ELIGIBILITY:
Inclusion Criteria:

* • Silicone oil (SO) tamponade ( up to 6 months)

  * Attached retina under SO
  * Attached retina 3 months after Silicone oil Removal (SOR)
  * Normal fellow eye ( no retinal detachment or macular disease)
  * OCT scan performed for the operated eyes (before SOR, and 3 months after SOR), and for the fellow eye (at any time during the study)

Exclusion Criteria:

* • Rhegmatogenous Retinal Detachment (RRD) with other tamponades ( e.g.: Gas, Densiron)

  * SO tamponade less than 3 months, or more than 6 months
  * Recurrent RD under SO
  * Recurrent RD within 3 months after SOR
  * One eyed
  * Vitrectomized fellow eye
  * Retinal detachment, or macular disease in the fellow eye.
  * Posterior staphyloma
  * Anisometropia (history, refraction if possible, spectacles prescription)
  * Absence of any of the OCT scans performed for the operated eyes (before SOR, and 3 months after SOR), and for the fellow eye (at any time during the study)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective Cohort study Retrospective review of records of eyes with Rhegmatogenous Retinal Detachment (RRD, for whom pars plana vitrectomy and silicone oil had been performed, in the period between January 2019 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Change in CFT just before SOR (central foveal thickness) | baseline to time just before silicone oil removal
  Change in CFT just before SOR (from baseline fellow eye) (microns, %) (each group)
Change in PFT just before SOR (Parafoveal thickness) | baseline to time just before silicone oil removal
  Change in PFT just before SOR (from baseline fellow eye) (microns, %) (each group)
• Change in CFT after SOR | from baseline fellow eye to 1 month after silicone oil removal
  • Change in CFT after SOR (from baseline fellow eye) (microns, %) (each group)
• Change in PFT after SOR | from baseline fellow eye to 1 month after silicone oil removal
  • Change in PFT after SOR (from baseline fellow eye) (microns, %) (each group)

SECONDARY OUTCOMES:
• Relative Risk of severe CFT Thinning before SOR (between group A and B) | baseline to time just before silicone oil removal
  • Relative Risk of severe CFT Thinning before SOR (between group A and B)
• Relative Risk of severe PFT Thinning before SOR (between group A and B | baseline to time just before silicone oil removal
  • Relative Risk of severe PFT Thinning before SOR (between group A and B
• Relative Risk of severe CFT Thinning after SOR (between group A and B) | from baseline fellow eye to 1 month after silicone oil removal
  • Relative Risk of severe CFT Thinning after SOR (between group A and B)
• Relative Risk of severe PFT Thinning after SOR (between group A and B) | from baseline fellow eye to 1 month after silicone oil removal
  • Relative Risk of severe PFT Thinning after SOR (between group A and B)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ewais WA, Ali LS, Aboalazayem FM. Impact of duration of silicone oil tamponade on foveal and parafoveal thickness in rhegmatogenous retinal detachment: a retrospective cohort study. Int Ophthalmol. 2024 Apr 2;44(1):167. doi: 10.1007/s10792-024-03096-8. PMID 38565753